CLINICAL TRIAL: NCT06130670
Title: Clinical Efficacy and Safety of Dexmedetomidine as an Adjuvant to Bupivacaine in Ultrasound-guided Quadratus Lumborum Versus Epidural Block for Postoperative Analgesia in Lower Abdominal Cancer Surgeries.
Brief Title: Clinical Efficacy and Safety of Dexmedetomidine as an Adjuvant in Quadratus Lumborum Versus Epidural Block in Postoperative Lower Abdominal Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Ahmed Hamed Mohamed, resident doctor/Demonstrator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: dexmedetomidine as an adjuvant
Record Dates: First submitted 2023-11-05; First posted 2023-11-14 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: To Compare Efficacy of Dexmedetomidine in Bilateral Quadratus Lumborum vs Lumbar Epidural Blocks on Analgesia After Major Lower Abdominal Surgery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Comparing the efficacy of Dexmedetomidine in bilateral quadratus lumborum block versus lumbar epidural block on postoperative analgesia following major lower abdominal cancer surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1:Ultrasound-guided quadratus lumborum block technique (Other): Ultrasound-guided quadratus lumborum block technique:
  the patients were placed in the lateral position. Following disinfecting of the site of injection, a convex probe (2-5 HZ, Edge, Sonosite, Seattle, the USA) was positioned in a parasagittal oblique plane at the L3-L4 level, which is approximately 4 cm from the posterior midline. The iliac crest, erector spinae (ES) muscle, QL muscle, and psoas (PM) muscle were identified, and a an 18-gauge Touhy's epidural needle (BBRAUN epidural set) was directed to the anterior part of the QL. Then, the needle tip was located between the QL and PM using the in-plane technique. Normal saline 5 mL was used to identify the plane. After confirmation of the injection site, 20 ml of 0.25% Bupivacaine bolus was injected and 1 μg/kg of dexmedetomidine dissolved in 2 ml normal saline were injected also between the QL and PM muscles divided equally on each side of the abdominal wall before induction general anesthesia.
  Interventions: Other: nerve block
- Group2:Lumbar epidural block (Other): Lumbar epidural block:
  Under strict aseptic precautions, lumbar epidural was performed for patients in Group II using a 16-gauge Touhy epidural needle by a median approach. The L3 - L4 interspaces was chosen for the injection. The epidural space identified by the loss of resistance technique. The catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of (3 mL) 2% lidocaine was given after the placement of the epidural catheter.
  In the epidural catheter a bolus dose of 15 ml bupivacaine 0.25% and 1 μg/kg of dexmedetomidine dissolved in 2 ml normal saline was injected before induction of general anesthesia.
  Interventions: Other: nerve block

INTERVENTIONS:
Other: nerve block — Comparing the efficacy of Dexmedetomidine in bilateral quadratus lumborum block versus lumbar epidural block on postoperative analgesia following major lower abdominal cancer surgery.

SUMMARY:
Clinical efficacy and safety of dexmedetomidine as an adjuvant in quadratus lumborum versus epidural block in postoperative patients

DETAILED DESCRIPTION:
One of the main concerns of patients presenting for major abdominal surgery and anesthesiologists who are involved in postoperative care is postoperative analgesia[1].

Despite improvements in surgical technique and perioperative care, complications in the immediate post-operative period remain significant [2]. The patients often experience significant post-operative pain and functional impairment and need 5-10 days to recover [3], [4].

Poor postoperative pain control leads to longer postoperative care, longer hospital stay and decreased patient overall satisfaction [5]. Opioids remain the mainstay of postoperative pain relief but have their own side effects. Therefore, the use of a multimodal analgesic strategy is nowadays preferable in most clinical settings to minimize the need for opioids. The use of regional anesthetic techniques provides excellent analgesia, as their effect can extend beyond the perioperative period [6].

As an important element of multimodal analgesia, regional blocks can reduce the dosage of opioids, minimize side effects, and enhance the quality of recovery after surgery [7].

Ultrasound-guided Quadratus Lumborum Block (QLB) is a relatively new regional anesthetic technique that was first described by Professor R. Blanco in 2007 at the annual scientific meeting of the European Society of Regional Anesthesia [8], it is relatively easily performed, the block effect lasts 24 - 48 h and up till now, no complications have been described during or after the block performance. QLB is safe and has found its place in multimodal postoperative pain strategy in patients undergoing abdominal surgery [9]. Quadratus lumborum block (QLB) is an emerging truncal block technique, [10] which includes injecting local anesthetic (LA) into the thoracolumbar fascia (TLF) surrounding the quadratus lumborum (QL) muscle. The analgesic effect is produced by the LA spreading along the TLF into the thoracic paravertebral space and transversalis fascia. QLB is an effective analgesic method for patients undergoing abdominal and hip surgeries [11,12 ,13 ,14]. Based on the different injection sites, there are four types of QLB, namely, lateral QLB, posterior QLB, transmuscular QLB, and intramuscular QLB. Transmuscular QLB includes the injection of LA between the QL muscle and the psoas major (PM) muscle. Transmuscular QLB can be implemented at the L4 and L2 levels using the subcostal approach [15]. Hesham et al. [16] have reported that the use of the subcostal approach to Transmuscular QLB can provide appropriate sensory blockade for open urological surgeries.

Epidural anesthesia is a technique for perioperative pain management with multiple applications in anesthesiology. It is useful as a primary anesthetic, but most commonly, it is used as a pain management adjuvant. It can be a single shot or a continuous infusion for long-term pain relief. Aside from the benefit of potentially providing excellent analgesia, its use reduces the exposure to other anesthetics and analgesics, decreasing side effects. It has also shown to decrease cortisol levels, expedite the return of bowel function, decrease the incidence of PE and DVT in the postoperative period, and shorten lengths of in-hospital stay.[17][18][19]

Regarding major lower abdominal surgery, epidural analgesia was shown to be the gold standard time-tested technique for providing postoperative analgesia, but due to its possible complications, contraindications, there is a need for other equally efficient analgesic techniques [20].

Adjuvant to local anesthetics is an evolving and exciting field of anesthesia practice with new technology promising to improve patient satisfaction and safety. While opioids continue to be the most commonly used local anesthetic adjuvant in clinical practice, alpha-2 receptor antagonists, especially dexmedetomidine, has been shown to potentiate the effect of local anaesthetics with an acceptable safety profile. Use of adjuvants to local anesthetic should take into consideration the available evidence and the advocated safe dose ranges, its effective routes of administration, the adverse effect profile of use of such adjuncts as well as preparedness to manage life threatening complications such as Local Anesthesia Systemic Toxicity (LAST). Its users should be aware of its neurotoxicity potential following perineural use and watch for its clinical implications. Search for newer molecules and techniques allowing for lesser perineural doses of local anesthetic, enhanced analgesic effect and improved safety profile are expected to guide further studies in future to fill up the present lacuna in evidence about the use of adjuvant for local anaesthetics.(21)

There are many adjuvants to local anesthesia that has been used in QLB and epidural analgesia such as: magnesium sulfate ,opioids ,dexamethasone,dexmedetomidine,etc.

The advantages of dexmedetomidine include reductions in cognitive dysfunction [22], respiratory depression [23, 24], ICU stays [25, 26], and financial costs [27]. Furthermore, it appears that dexmedetomidine can act synergistically when used in conjunction with other analgesic or anesthetic medications and can reduce their side effects [28-30]. However, it has been suggested that dexmedetomidine reduces both heart rate [31] and blood pressure [24].

The addition of dexmedetomidine to other anesthetic agents during epidural procedures provided a longer duration of analgesia, as well as highly significant improvements in the time to sensory block and the sedation score, and decreased the requirement for rescue analgesia.(32) Interfascial dexmedetomidine adjuvant to QLB provided better postoperative analgesia in terms of less morphine consumption, better pain scores and longer time to first analgesic request when compared with the IV dexmedetomidine.(33) In this study we will compare the effect of dexmedetomidine in bilateral quadratus lumborum block and lumbar epidural block on postoperative analgesia.

Aim(s) of the Research :

Comparing the efficacy of Dexmedetomidine in bilateral quadratus lumborum block versus lumbar epidural block on postoperative analgesia following major lower abdominal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patient's 18-70years old
2. ASA I-II and NYHA I-II.
3. type of surgery: major lower abdominal cancer surgery

Exclusion Criteria:

1. Patients who refused to participate in the study.
2. coagulation disorders.
3. opioid dependence.
4. sepsis or local infection at or near the vicinity of the block site.
5. patients with psychiatric illnesses that would interfere with perception and assessment of pain.
6. allergy to any of the studied drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | the first 24 hrs after surgery
  Time of first analgesic request during the first 24 hrs after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Xu W, Daneshmand S, Bazargani ST, Cai J, Miranda G, Schuckman AK, Djaladat H. Postoperative Pain Management after Radical Cystectomy: Comparing Traditional versus Enhanced Recovery Protocol Pathway. J Urol. 2015 Nov;194(5):1209-13. doi: 10.1016/j.juro.2015.05.083. Epub 2015 Aug 13. PMID 26021824
- [Background] Patel HD, Ball MW, Cohen JE, Kates M, Pierorazio PM, Allaf ME. Morbidity of urologic surgical procedures: an analysis of rates, risk factors, and outcomes. Urology. 2015 Mar;85(3):552-9. doi: 10.1016/j.urology.2014.11.034. PMID 25733265
- [Background] Bhalla RG, Wang L, Chang SS, Tyson MD. Association between Preoperative Albumin Levels and Length of Stay after Radical Cystectomy. J Urol. 2017 Nov;198(5):1039-1045. doi: 10.1016/j.juro.2017.05.066. Epub 2017 May 19. PMID 28533006